CLINICAL TRIAL: NCT00433836
Title: A Multicenter, Randomized, Double-blind, Parallel-group, Evaluation of 12 Weeks of Valsartan Compared to Enalapril on Sitting Systolic Blood Pressure in Children 6 to 17 Years of Age With Hypertension
Brief Title: Effect of Valsartan Compared to Enalapril on Sitting Systolic Blood Pressure in Children With High Blood Pressure
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: External Affairs, Novartis Pharmaceuticals
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CVAL489K2302
Record Dates: First submitted 2007-02-08; First posted 2007-02-12 (Estimated); Results first posted 2011-05-19 (Estimated); Last update posted 2011-05-19 (Estimated); Status verified 2011-04

CONDITIONS: Hypertension
Keywords: Children; pediatrics; High Blood Pressure; Hypertension; Valsartan; enalapril
MeSH Terms: conditions — Hypertension | interventions — Valsartan; Enalapril

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator

ARMS (6):
- Valsartan 80 mg (Experimental)
  Interventions: Drug: Valsartan
- Valsartan 160 mg (Experimental)
  Interventions: Drug: Valsartan
- Valsartan 320 mg (Experimental)
  Interventions: Drug: Valsartan
- Enalapril 10 mg (Active Comparator)
  Interventions: Drug: Enalapril
- Enalapril 20 mg (Active Comparator)
  Interventions: Drug: Enalapril
- Enalapril 40 mg (Active Comparator)
  Interventions: Drug: Enalapril

INTERVENTIONS:
Drug: Valsartan — Weight stratified dosages given by mouth, once daily, of valsartan 80/160/320 mg.
  Arms: Valsartan 160 mg; Valsartan 320 mg; Valsartan 80 mg
Drug: Enalapril — Weight stratified dosages given by mouth, once daily, of enalapril 10/20/40 mg.
  Arms: Enalapril 10 mg; Enalapril 20 mg; Enalapril 40 mg

SUMMARY:
The purpose of this 12-week active controlled trial is to evaluate the safety and efficacy of valsartan 80/160/320 mg (weight stratified) compared with enalapril 10/20/40 mg (weight stratified) on sitting systolic blood pressure (SSBP) in 6 - 17 year old children with hypertension (SSBP ≥ 95th percentile for age gender and height).

ELIGIBILITY:
Inclusion Criteria:

* Male or female, ages 6-17, with a documented history of hypertension
* Must be able to swallow a pill
* Must be ≥ 18 kg or ≤160 kg
* MSSBP (mean of 3 measurements) must be ≥ 95th percentile, for age, gender and height, at Visit 2 (randomization), by office blood pressure measurement
* Patients who are eligible and able to participate in the study and whose parent(s)/guardian(s) consent in writing (written informed consent) to their doing so after the purpose and nature of the investigation has been clearly explained to them. (An assent will be required for some patients depending upon their age and local requirements regarding assents)

Exclusion Criteria:

* Renal artery stenosis
* Current diagnosis of heart failure (NYHA Class II-IV).
* MSSBP ≥ 25% above the 95th percentile
* Second or third degree heart block without a pacemaker.
* Concurrent potentially life threatening arrhythmia or symptomatic arrhythmia.
* Clinically significant valvular heart disease.
* Patient that demonstrates clinically significant ECG abnormalities other than those associated with left ventricular hypertrophy.
* Previous solid organ transplantation except renal, liver or heart transplantation. Renal, liver or heart transplant must have occurred at least 6 months prior to enrollment. Patient must be on stable doses of immunosuppressive therapy for 3 months and deemed clinically stable by the investigator.

Other protocol-defined inclusion/exclusion criteria may apply

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Actual)
Dates: Start 2007-01; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (11):
- Sites in USA, East Hanover, New Jersey, United States
- Sites in Belgium, Sites in Belgium, Belgium
- Sites in France, Sites in France, France
- Sites in Germany, Sites in Germany, Germany
- Sites in Hungary, Hungary, Hungary
- Sites in India, Sites in India, India
- Sites in Italy, Sites in Italy, Italy
- Sites in Poland, Poland, Poland
- Sites in Slovakia, Slovakia, Slovakia
- Sites in Sweden, Sites in Sweden, Sweden
- Sites in Turkey, Turkey, Turkey (Türkiye)

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Valsartan | Enalapril
Started | 151 | 149
Completed | 138 | 143
Not Completed | 13 | 6
Not completed — Adverse Event | 7 | 0
Not completed — Lost to Follow-up | 3 | 0
Not completed — Withdrawal by Subject | 2 | 1
Not completed — Unsatisfactory therapeutic effect | 1 | 1
Not completed — Protocol Violation | 0 | 2
Not completed — Condition no longer requires study drug | 0 | 1
Not completed — Abnormal laboratory values | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Valsartan | Enalapril | Total
Number analyzed (Participants) | 151 | 149 | 300
Age Continuous [Mean (Standard Deviation); unit: years] | 12.7 (2.93) | 13.0 (2.94) | 12.9 (2.93)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 44 | 109
  Male | 86 | 105 | 191

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Mean Sitting Systolic Blood Pressure (MSSBP)
Description: Mean sitting systolic blood pressure (MSSBP) change after 12 weeks of treatment measured by office blood pressure measurement.
Time Frame: Baseline and Week 12
Population: Intent-to-treat. Only patients who had both baseline and endpoint values are included.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Valsartan | Enalapril
Number analyzed (Participants) | 148 | 148
mm Hg | -15.4 (1.29) | -14.1 (1.28)
Statistical Analysis 1: Comparison: Valsartan vs Enalapril; Test type: Non-Inferiority or Equivalence — non-inferiority delta of 3.5 mm Hg; ANOVA; Mean Difference (Final Values) = -1.3, 95% CI 2-sided [-3.80 to 1.17]

2. Secondary Outcome: Change From Baseline in Mean Sitting Diastolic Blood Pressure (MSDBP)
Description: The change from baseline in mean sitting diastolic blood pressure (MSDBP) after 12 weeks of treatment as measured by office blood pressure.
Time Frame: Baseline and Week 12
Population: Intent-to-treat. Only patients who had both baseline and endpoint values are included.
Measure: Least Squares Mean (Standard Error); unit: mm Hg
Arm/Group | Valsartan | Enalapril
Number analyzed (Participants) | 148 | 148
mm Hg | -9.4 (0.94) | -8.5 (0.95)

3. Secondary Outcome: Decrease in MSSBP to < 95th Percentile for Age, Gender and Height
Description: The percentage of children whose MSSBP decreased to <95th percentile for age, gender, and height on valsartan vs. enalapril monotherapy at week 12.
Time Frame: at week 12
Population: Intent-to-treat. Only patients who had both baseline and endpoint values are included.
Measure: Number; unit: Percentage of participants
Arm/Group | Valsartan | Enalapril
Number analyzed (Participants) | 148 | 148
Percentage of participants | 66.9 | 70.3

4. Secondary Outcome: Change From Baseline in Mean Ambulatory Systolic Blood Pressure (ASBP) and Mean Ambulatory Diastolic Blood Pressure (ADBP) Over 24 Hours in Subset of Patients
Description: The effect of valsartan and enalapril between baseline and visit 6 on 24-hour mean ambulatory systolic and diastolic blood pressure (ASBP, ADBP) in a subset of patients.
Time Frame: Baseline and Week 8
Population: A subset of approximately 100 - 150 patients from selected centers was expected to undergo Ambulatory Blood Pressure Monitoring at baseline (Week 0) and at Week 8; however, only 56 patients chose to participate in this aspect of the study.
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Valsartan | Enalapril
Number analyzed (Participants) | 26 | 30
mm Hg
  ASBP | -9.8 (6.75) | -6.8 (7.41)
  ADBP | -9.3 (6.27) | -5.5 (5.73)

ADVERSE EVENTS:
Description: Includes all patients who received at least one dose of post-randomization study drug; patients were analyzed according to the actual treatment received.
Arm/Group | Valsartan | Enalapril
Serious Adverse Events (participants affected / at risk) | 3/151 | 2/148
Other Adverse Events (participants affected / at risk) | 42/151 | 52/148
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan (N=151) | Enalapril (N=148)
Avulsion fracture (Injury, poisoning and procedural complications) | 0 | 1
Renal injury (Injury, poisoning and procedural complications) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Brain injury (Nervous system disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Valsartan (N=151) | Enalapril (N=148)
Nasopharyngitis (Infections and infestations) | 10 | 8
Pharyngitis (Infections and infestations) | 6 | 11
Upper respiratory tract infection (Infections and infestations) | 10 | 7
Headache (Nervous system disorders) | 18 | 28
Cough (Respiratory, thoracic and mediastinal disorders) | 9 | 10

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.